## Cover Page Evaluation of the Effect of Intravitreal Injections of Anti-VEGF on Macular Perfusion in Diabetic Patients Using OCTA (IMPACT) NCT03246152

**Document date: 5/16/2019** 

**Upload date: 1/13/2020** 

## **Statistical methods:**

Data were coded and entered using the statistical package SPSS (Statistical Package for the Social Sciences) version 25. Data was summarized using mean, standard deviation, median, minimum and maximum in quantitative data and using frequency (count) and relative frequency (percentage) for categorical data. Comparisons between quantitative variables were done using the non-parametric Kruskal-Wallis and Mann-Whitney tests. For comparison of serial measurements within same patients paired t test was used in normally distributed quantitative variables while non-parametric Wilcoxon signed rank test was used for distributed quantitative variables non-normally (Chan, 2003a). Correlations between quantitative variables were done using Pearson or Spearman correlation coefficient (Chan, 2003b). Linear regression analysis was done to predict changes in different parameters using baseline data *(Chan, 2004)*. P-values less than 0.05 were considered as statistically significant.

## Ref:-

**Chan YH (2003a):** Biostatistics102: Quantitative Data – Parametric & Non-parametric Tests. Singapore Med J.;44(8): 391-396.

**Chan YH (2003b):** Biostatistics 104: Correlational Analysis. Singapore Med J.;44(12): 614-619.

**Chan YH (2004):** Biostatistics 201: linear regression analysis. Singapore Med J.;45(2): 55-61.